CLINICAL TRIAL: NCT05779150
Title: Efficacy of CeraVe® Moisturizing Cream on Skin Pruritus in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2023-004
Record Dates: First submitted 2023-03-04; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: self-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): Routine treatment together with once applicating CeraVe® Moisturising Cream after daily bath.
  Interventions: Other: CeraVe® Moisturising Cream
- Control Group (Placebo Comparator): Routine treatment together with once applicating Standard Cream after daily bath.
  Interventions: Other: Standard Cream

INTERVENTIONS:
Other: CeraVe® Moisturising Cream — CeraVe® Moisturising Cream contains 3 kinds of skin-native ceramides, which can protect the skin against external stimuli, strengthen the damaged skin barrier, fill the intercellular lipids to deeply trap water, relieve dry skin, and increase skin hydration.
  Arms: Case group
Other: Standard Cream — placebo cream
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate the CeraVe® moisturizing cream's efficiency on the improvement of skin barrier in patients with chronic elderly pruritus. The main questions it aims to answer are:

type of study: clinical trial participant population:in patients with chronic elderly pruritus [question 1] Evaluate the CeraVe® moisturizing cream's efficiency on the improvement of skin barrier in patients with chronic elderly pruritus, including improvements of redness, dryness/squamation, itching, burning, tingling, tightness and other factors.

[question 2] Evaluate the tolerance of CeraVe® Moisturising Cream. [question 3] Evaluate the product experience of patients who were utilizing CeraVe® Moisturising Cream.

This trial utilizing simple randomization, the left and right calves of paticipants were randomly divided into test side(applicating CeraVe® Moisturising Cream ) and control side (applicating Standard Cream)according to random number representation. Grouping results were double-blinded.

ELIGIBILITY:
Inclusion Criteria:

* patients age≥60 years old(male or female).
* Clinician evaluates dry pruritus or patient complains of pruritus, which lasts for more than 1 month.
* Patients informed consent to the purpose and content of the research, willing to cooperate with follow-up observation. Have good communication and understanding skills.
* Patients are willing to share photos for medical research purpose.

Exclusion Criteria:

* Patients with bacterial and/or viral infections in the acute phase of skin inflammation
* The affected area is complicated by other skin diseases that may affect the efficacy evaluation
* Those who are allergic to the ingredients of this product or with allergic constitution
* Patients who have severe heart, brain, lung, or liver damage.
* Those who have received systemic or local antiallergic drug treatment within 2 weeks before enrollment of this study.
* Those who attending other clinical drug trials within 4 weeks before enrollment of this study.
* Patients with a history of alcohol or drug abuse.
* Patients who are unwilling to sign the informed consent form, and those who are unwilling to cooperate.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-26 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-02-03 (Estimated)

PRIMARY OUTCOMES:
change from baseline effective rate of treatment at 14 days after treatment | baseline and 14 days after treatment
  1. According to Nimodipine calculation: Treatment Index = (Self-assessment parameters after treatment - Self-assessment parameters before treatment)/Self-assessment parameters before treatment*100%
  2. Definition:
     Cure: No symptoms, Treatment index > 95% Significant Recovery: symptoms are significantly relieved, 70% <Treatment index≤95% Improved: Symptoms improved, 30%≤Treatment index≤70% No effect: No change in symptoms, Treatment index <30%
  3. Effective rate of treatment = (Cure + Significant recovery)/total*100%

SECONDARY OUTCOMES:
clinical tolerability score | 1 day, 3 days, 7 days, and 14 days after treatment
  The clinical tolerability score mainly evaluates the objective parameters and subjective parameters.
  Objective parameters include rash, edema, redness, dryness/desquamation, desquamation, and other superficial signs, and each individual item is scored on a scale of 0 to 3 (level 0 is none, level 1 is slight, level 2 is obvious, level 3 is serious ); Subjective parameters include burning, tingling, itching, tightness, tingling, and other Follow upnctional manifestations, and each individual item is scored on a scale of 0 to 3 (level 0 is none, level 1 is slight, level 2 is obvious, level 3 level is serious); The clinical tolerability score is the average of objective parameters and subjective parameters, which is calculated by the sum of 6 objective parameters and 6 subjective parameters divided by 12.
product experience score | after 14 days of treatment
  the evaluation includes: improvement in overall skin appearance, product's texture, convenience of product, applicating texture, product's envelopment, product's absorption, product's rub feeling on skin, product's gentleness on skin, product's comfort on skin, product's greasy feeling, product's suitable for skin, product's overall delight, those 12 aspects will be express on 1-5 score scale(1: Completely Disagree; 2:Somewhat disagree;3:neither agree nor disagree;4:somewhat agree;5:completely Agree). The product experience score is the average of those 12 aspects, calculate by the sum of 12 aspects rating divided by 12.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hu, Dr, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No